CLINICAL TRIAL: NCT03030313
Title: Assessment of the Temporal Changes in Nightly Respiration Rate in Combination With a Daily Symptom Reporting Application for Facilitating Early Treatment of Symptoms in COPD Patients
Brief Title: Respiration Rate Monitoring in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MA-16-05-01
Record Dates: First submitted 2016-11-18; First posted 2017-01-25 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respiration rate monitoring (Experimental): Reassure Non-Contact Respiration Monitor
  Interventions: Device: Reassure Non-Contact Respiration Monitor

INTERVENTIONS:
Device: Reassure Non-Contact Respiration Monitor — Reassure Respiration Monitor uses very low power radio waves to detect respiratory movements of a person while asleep in bed - without physical contact with the individual. Algorithms analyze the respiratory movement signals and extract information about respiration rate and variability. This data is uploaded to a secure cloud infrastructure for storage.

SUMMARY:
Assess the feasibility of using remote respiration rate monitoring as a component of home care, how respiration rate data may be used in combination with other data to potentially improve response to symptoms, and to generate data to inform the endpoints and effect sizes of future studies.

DETAILED DESCRIPTION:
The research question is whether monitoring of respiration rates and variability can be helpful in management of COPD patients in conjunction with or separately from self-reported symptom scores using the COPD Co-PILOT application. Current techniques (such as patient's self-reported symptoms) have limited sensitivity and specificity with regard to predicting decompensation. Measurement of respiration parameters and the variability of the parameters may detect worsening COPD. Changes in respiration patterns may occur sufficiently far in advance of decompensation (e.g. >5 days prior to patient symptoms) such that it would allow an opportunity for earlier intervention with medical assessment and current therapeutic approaches.

The specific primary aim includes evaluation of the correlation of respiration rate parameters to indicators of healthcare utilization including drug changes, office or ER visits, hospitalization, or other clinical interventions. Secondary aims include evaluation of (i) the sensitivity and specificity of respiration rate monitoring results to predict COPD worsening requiring medical intervention, (ii) the sensitivity and specificity of respiration rate monitoring results in conjunction with COPD Co-PILOT scores or components to predict COPD worsening requiring medical intervention, and the correlation of respiration rate parameters to episode duration as defined by number of days from COPD Co-PILOT Score >1 to resolution (COPD Co-PILOT Score <1 for 7 consecutive days).

ELIGIBILITY:
Inclusion Criteria:

* Males or females age ≥35 years old
* Documented diagnosis of moderate to very severe COPD (GOLD Level II-IV)
* Weight ≥35 kg
* Currently using the COPD Co-PILOT application (at least 3 months with 70% compliance)
* Must be able to read and understand English and consent for themselves

Exclusion Criteria:

* Currently using any form of non-invasive positive airway pressure ventilation
* Diagnosis of significant heart failure (NYHA Class III or IV)
* Cognitive impairment (determined by physician) that will make it hard to follow instructions regarding device usage
* BMI ≥45.5
* Residing in hospice care, Skilled Nursing Facilities or Long Term Acute Care facilities
* Currently using a wearable drug infusion pump to deliver medication
* Planned procedures at time of enrollment that will occur within timeframe of study and require hospitalization etc.
* Declines to participate at any time.
* In the opinion of the Investigator, may be non-compliant with study schedules or procedures
* No cellular coverage at their primary residence

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Correlation of Respiration Rate to Indicators of Healthcare Utilization | 12 weeks
  Indicators of healthcare utilization include change in medications for COPD, number of office or ER visits, number of hospitalizations.

SECONDARY OUTCOMES:
Sensitivity and Specificity of Respiration Rate to Predict COPD Worsening | Baseline to 12 weeks
Sensitivity and Specificity of Respiration Rate in Conjunction with COPD Co-PILOT Scores to Predict COPD Worsening | 12 weeks
Correlation of Respiration Rate to COPD Episode Duration | 12 weeks
  Episode duration is defined by number of days from COPD Co-PILOT Score >1 to resolution (COPD Co-PILOT Score <1 for 7 consecutive days)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Criner, MD, Principal Investigator — Temple University
Locations (1):
- HGE Health Care Solutions, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No